CLINICAL TRIAL: NCT02456194
Title: Management of Traumatic Bone Defects in Tibial Plateau Fractures With Antibiotic-Impregnated Biodegradable Calcium Sulfate Beads: A Prospective Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ross Leighton (Other)
Collaborators: Biocomposites Ltd (Industry)
Responsible Party: Sponsor-Investigator, Ross Leighton, Orthopaedic Surgeon, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RL007
Record Dates: First submitted 2015-05-26; First posted 2015-05-28 (Estimated); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2022-11

CONDITIONS: Tibial Fractures; Intra-Articular Fractures; Fracture Fixation, Internal
MeSH Terms: conditions — Tibial Fractures; Intra-Articular Fractures | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Calcium Sulfate + Antibiotics + Internal Fixation (Experimental)
  Interventions: Device: Calcium Sulfate + Antibiotics + Internal Fixation

INTERVENTIONS:
Device: Calcium Sulfate + Antibiotics + Internal Fixation — STIMULAN Rapid Cure, mixed with antibiotic, and prepared in bead form. Must be used in conjunction with internal fixation. Choice of antibiotic is left to the surgeon's discretion.
  Other Names: STIMULAN Rapid Cure

SUMMARY:
This is a prospective clinical trial of tibial plateau fractures treated with internal fixation and a calcium sulfate graft which can be mixed with antibiotics and molded into various bead sizes for implantation into bone defects. The graft material chosen for this study is STIMULAN Rapid Cure (Biocomposites, UK), which is approved for use as a bone void filler and may be mixed with a variety of antibiotics. The combination of STIMULAN + antibiotic in bead form is the "study device".

Our primary study aim is to look at resorption and remodeling of the study device into bone. Another important aim of the study is to look at subsidence, or collapse, of the joint surface.

ELIGIBILITY:
Inclusion Criteria:

* Adult (skeletally mature) men or women;
* Acute, closed, tibial plateau fractures, Schatzker grade 1 through 5;
* Internal fixation and use of study device per protocol;
* Fracture repair within 30 days of injury;
* Signed informed consent to participate in study.

Exclusion Criteria:

* Uncontrolled diabetes;
* Severe degenerative or metabolic bone disease;
* Malignancy;
* Severe vascular or neurologic disease;
* Alcoholism;
* Substance abuse;
* Use of systemic steroids;
* Immunosuppressive therapy;
* Hypercalcaemia;
* Renal-compromised patients;
* Osteomyelitis or chronic infection in the study limb;
* Women who are pregnant or breast-feeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09; Primary Completion 2019-04 (Actual); Study Completion 2021-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ross Leighton, MD, Principal Investigator — Nova Scotia Health Authority
Locations (5):
- Canada (5):
  - Alberta Health Services, Calgary, Alberta
  - Horizon Health Network, Moncton, New Brunswick
  - Memorial University of Newfoundland, St. John's, Newfoundland and Labrador
  - Halifax Infirmary, Halifax, Nova Scotia
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Started | 30
Completed | 29
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 30

OUTCOME MEASURES:

1. Primary Outcome: Resorption of Study Device
Description: Number of participants with any study device remaining visible on CT
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
Participants | 4

2. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Pain Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
score on a scale | 89.0 (18.6)

3. Secondary Outcome: Range of Motion
Description: Range of knee motion (active flexion) in degrees
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 26
degrees | 97.38 (27.42)

4. Secondary Outcome: Subsidence of Joint Surface
Description: Amount of collapse of the joint surface, measured in mm, on plain x-ray. Reported as number of participants with at least 2mm of subsidence on x-ray.
Time Frame: 6 weeks, 3 months, 6 months, 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
Participants | 4

5. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Pain Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
score on a scale | 51.71729611 (23.47939809)

6. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Pain Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
score on a scale | 62.18 (23.07)

7. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Pain Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
score on a scale | 70.21 (21.76)

8. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Pain Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 29
score on a scale | 75.38 (19.60)

9. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Symptoms Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
score on a scale | 89.29 (14.85)

10. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Symptoms Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
score on a scale | 55.79 (20.63)

11. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Symptoms Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
score on a scale | 62.86 (23.32)

12. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Symptoms Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
score on a scale | 57.98 (22.44)

13. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Symptoms Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 29
score on a scale | 70.69 (18.37)

14. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Activities of Daily Living Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
score on a scale | 92.24 (17.00)

15. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Activities of Daily Living Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
score on a scale | 50.37 (23.92)

16. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Activities of Daily Living Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
score on a scale | 67.42 (21.98)

17. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Activities of Daily Living Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
score on a scale | 74.54 (19.45)

18. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Activities of Daily Living Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 29
score on a scale | 81.68 (16.51)

19. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Sports/Recreation Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
score on a scale | 81.9 (28.5)

20. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Sports/Recreation Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
score on a scale | 14.62 (29.81)

21. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Sports/Recreation Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
score on a scale | 22.93 (22.12)

22. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Sports/Recreation Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
score on a scale | 39.17 (35.78)

23. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Sports/Recreation Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 29
score on a scale | 53.5 (28.49)

24. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Quality of Life Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
score on a scale | 85.34 (26.8)

25. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Quality of Life Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
score on a scale | 25 (22.46)

26. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Quality of Life Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
score on a scale | 35.83 (23.93)

27. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Quality of Life Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
score on a scale | 46.04 (27.07)

28. Secondary Outcome: Knee Injury Osteoarthritis Outcome Score - Quality of Life Subscale
Description: Self-reported outcome score, reported as the mean score at each time point. Scale 0-100, 100 is best.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 29
score on a scale | 58.98 (23.47)

29. Secondary Outcome: Range of Motion
Description: Range of knee motion (active flexion) in degrees
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 27
degrees | 108.52 (25.35)

30. Secondary Outcome: Range of Motion
Description: Range of knee motion (active flexion) in degrees
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 29
degrees | 121.20 (19.98)

31. Secondary Outcome: Range of Motion
Description: Range of knee motion (active flexion) in degrees
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 29
degrees | 126.51 (11.87)

32. Secondary Outcome: Resorption of Study Device
Description: Number of participants with any study device remaining visible on x-ray
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 29
Participants | 8

33. Secondary Outcome: Resorption of Study Device
Description: Number of participants with any study device remaining visible on x-ray
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
Participants | 4

34. Secondary Outcome: Resorption of Study Device
Description: Number of participants with any study device remaining visible on x-ray
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
Number analyzed (Participants) | 30
Participants | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Calcium Sulfate + Antibiotics + Internal Fixation
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 6/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Calcium Sulfate + Antibiotics + Internal Fixation (N=30)
articular surface apoptosis (Musculoskeletal and connective tissue disorders) | 1 — Theparticipant had healed their fracture by three months but had articular surface apoptosis by six months following the initial fracture and was revised to a total knee replacement at nine months and went on to heal uneventfully.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Calcium Sulfate + Antibiotics + Internal Fixation (N=30)
Infection (Infections and infestations) | 2 — Treated with irrigation and debridement and antibiotics
intra-articular heterotopic bone formation (Musculoskeletal and connective tissue disorders) | 1 — debrided arthroscopically
hardware irritation (Musculoskeletal and connective tissue disorders) | 3 — treated with revision to smaller plate or removal

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-03-31): https://cdn.clinicaltrials.gov/large-docs/94/NCT02456194/Prot_SAP_000.pdf
  • Informed Consent Form (2015-07-16): https://cdn.clinicaltrials.gov/large-docs/94/NCT02456194/ICF_001.pdf